CLINICAL TRIAL: NCT00369395
Title: A Phase 2, Open-Label, Two-Stage Study of Volociximab (M200) for the Treatment of Subjects With Metastatic Melanoma
Brief Title: A Study of Volociximab in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient clinical activity
Sponsor: Abbott (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206-MM-201
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Stage IV Melanoma
Keywords: melanoma; antibody; angiogenesis; volociximab
MeSH Terms: conditions — Melanoma | interventions — volociximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volociximab (Experimental): Volociximab 15 mg/kg
  Interventions: Drug: volociximab

INTERVENTIONS:
Drug: volociximab — Volociximab, 15 mg/kg, IV infusion once a week for 8 weeks. Subjects who achieved SD or better at Day 50 ± 2 days (Week 8) were eligible to continue receiving weekly infusions of volociximab until disease progression.

SUMMARY:
This is a Phase 2, multicenter, research study determining the effects of an investigational drug called volociximab in metastatic melanoma.

The purpose of the study is to compare the clinical benefit and safety of volociximab. Pharmacokinetics and mechanism of action will also be evaluated.

ELIGIBILITY:
Inclusion Criteria

1. Must give written informed consent and any authorizations required by local law (e.g., Protected Health Information [PHI]).
2. Aged >=18 years old at the time of informed consent.
3. Stage III and Stage IV unresectable melanoma with documented progression during or following the most recent prior melanoma therapy.
4. Must have failed at least 1 prior therapy for metastatic disease.
5. Must have at least 2 cutaneous, subcutaneous, or nodal metastases that are safely accessible for pre treatment and post treatment biopsies.
6. Must agree to pre-treatment and post-treatment biopsies of tumor lesions (subjects in Stage 1 only).
7. Must have at least 1 measurable target lesion for CT/MRI assessment, according to RECIST criteria.
8. ECOG Performance Status <=1.
9. Acceptable laboratory results
10. Life expectancy >=12 weeks.
11. Male subjects and female subjects of child bearing potential must be willing to practice effective contraception during the study and be willing and able to continue contraception for 4 months after last infusion of study treatment.

Exclusion Criteria

1. Subjects with any other active malignancy in addition to metastatic melanoma.
2. CNS metastases, unless stable for at least 2 months following definitive local therapy (surgery, stereotactic radiation). Subjects may not require treatment with steroids or anticonvulsants.
3. History of any other significant medical condition, including cardiovascular, pulmonary, neurologic, or autoimmune disease; active infections (e.g., bacterial or fungal); or a psychiatric condition within 6 months of Day 1
4. History of hepatitis B or C.
5. Known history of HIV infection or AIDS.
6. History of thromboembolic or cerebrovascular events, such as stroke, transient ischemic attack, deep vein thrombosis, or bleeding disorders within 12 months prior to Day 1.
7. Prior radiation therapy, chemotherapy, hormonal therapy, or immunotherapy for melanoma within 4 weeks prior to Day 1.
8. Previous exposure to volociximab.
9. Aspirin, high dose warfarin, or heparin use. (Note: Aspirin <=81 mg/day, low-dose warfarin 1 mg/day or low-dose heparin for IV catheter patency is allowed.)
10. Major surgery within 4 weeks prior to Day 1.
11. Requirement for immunosuppression, and/or systemic steroid therapy.
12. Investigational therapies within 4 weeks prior to Day 1 or 4 half lives of the prior investigational drug (whichever is longer).
13. Known hypersensitivity to murine or chimeric antibodies.
14. Any condition that, in the opinion of the Investigator, makes the subject unsuitable for study participation.
15. Female subjects who are pregnant or currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate at the Week 8 visit, defined as the number of subjects who have not progressed by the Week 8 visit | 8 weeks intervals

SECONDARY OUTCOMES:
Pharmacokinetics of volociximab | Every infusion and follow up visit
Assess safety by recording and evaluating adverse events (AEs); changes in vital signs, hematology, blood chemistry, and urinalysis parameters; and anti-volociximab antibody formation | Throught study and follow up period,approx. 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — Abbott
Locations (7):
- United States (7):
  - Site Reference ID/Investigator# 70357, Scottsdale, Arizona
  - Site Reference ID/Investigator# 70356, La Jolla, California
  - Site Reference ID/Investigator# 70375, Aurora, Colorado
  - Site Reference ID/Investigator# 70376, Boston, Massachusetts
  - Site Reference ID/Investigator# 70359, St Louis, Missouri
  - Site Reference ID/Investigator# 70380, Greenville, South Carolina
  - Site Reference ID/Investigator# 70377, Dallas, Texas